CLINICAL TRIAL: NCT01402869
Title: Methemoglobin Levels in Generally Anesthetized Pediatric Dental Patients Receiving Prilocaine Versus Lidocaine
Brief Title: Methemoglobin Levels in Generally Anesthetized Pediatric Dental Patients Receiving Local Anesthetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Lauren GutenBerg, Pediatric Dental Resident, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 5110172
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Results first posted 2014-04-25 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-03

CONDITIONS: Methemoglobinemia
Keywords: Methemoglobin; Methemoglobinemia; Prilocaine; Lidocaine
MeSH Terms: conditions — Methemoglobinemia | interventions — Prilocaine; Lidocaine; Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Prilocaine (Experimental): 30 subjects will receive 5mg/kg of 4% prilocaine plain local anesthetic for restorative dental treatment under general anesthesia
  Interventions: Drug: 4% prilocaine plain
- Lidocaine (Experimental): 30 subjects will receive 2.5mg/kg of 2% lidocaine with 1:100,000 epinephrine local anesthetic for restorative dental treatment under general anesthesia
  Interventions: Drug: 2% Lidocaine with 1:100,000 epinephrine
- No local anesthetic (No Intervention): 30 subjects will not receive local anesthetic for dental treatment under general anesthesia-Negative control

INTERVENTIONS:
Drug: 4% prilocaine plain — 5mg/kg via infiltration into multiple sites of the buccal mucosa of mouth 1 time prior to start of restorative dental treatment
  Other Names: Citanest Plain
  Arms: Prilocaine
Drug: 2% Lidocaine with 1:100,000 epinephrine — 2.5mg/kg via infiltration into multiple sites of buccal mucosa of mouth 1 time prior to restorative dental treatment
  Other Names: Xylocaine
  Arms: Lidocaine

SUMMARY:
To establish and compare maximum methemoglobin blood levels and times to maximum methemoglobin blood levels following the administration of the injectable local anesthetics prilocaine and lidocaine when used for dental treatment in pediatric patients under general anesthesia. Patients will be randomized into three equal study groups. Two of the study groups will receive local anesthetic and the third group will not. Methemoglobin blood levels will be non-invasively monitored and recorded throughout dental treatment for all groups using a Masimo Radical-7 Pulse Co-Oximeter device.

DETAILED DESCRIPTION:
Methemoglobin is an abnormal hemoglobin that is formed by the oxidation of one or more of the four heme groups of hemoglobin by oxygen and other exogenous oxidizing agents. The injectable local anesthetic prilocaine that is routinely used in the medical and dental professions is a well known inducer of methemoglobin. The injectable local anesthetic lidocaine has also been suggested to be associated with the development of methemoglobin; however, there is no direct evidence supporting these claims.

The concern with methemoglobin is that it is a dose-dependent toxin. The oxidation of one of the iron groups from a ferrous state to a ferric state alters the molecular structure of the hemoglobin molecule and impairs its ability to bind oxygen. This ultimately results in less oxygen being delivered to peripheral tissues and less carbon dioxide being removed which can cause tissue hypoxia. A small amount (0-2%) of methemoglobin is normally present in the blood as a result of the oxidation of hemoglobin by the prototypical oxidant oxygen. However, when an individual is exposed to an exogenous oxidizing agent of sufficient dosage and potency, methemoglobin levels can rise above 2% and a person can develop what is known as acquired methemoglobinemia. Signs of cyanosis as a result of acquired methemoglobinemia usually become present when methemoglobin blood levels rise above 15%.

Despite the injectable local anesthetic prilocaine being a well known inducer of methemoglobin and lidocaine being a speculated inducer, there are no documented studies or trials in the dental literature as to the extent of the amount of methemoglobin that is formed following the routine use of these injectable local anesthetics.

This investigation will examine the peak blood levels of methemoglobin and the time to the peak levels of methemoglobin following the use of injectable prilocaine and lidocaine when used for dental treatment in pediatric patients under general anesthesia.

This study population will consist of 90 patients, 3 to 6 years of age, scheduled to undergo comprehensive dental rehabilitation under general anesthesia at the Koppel Special Care Dentistry Center at Loma Linda University School of Dentistry. Following enrollment, subjects will be randomized into three equal study groups: 1) 4% prilocaine plain, 2) 2% lidocaine with 1:100,000 epinephrine, and 3) No local anesthetic. All subjects will have a Masimo Radical-7 pediatric, non-disposable, pulse co-oximeter sensor placed on the ring finger of the right hand following the induction of general anesthesia. The sensor will then be connected to a Radical-7 Pulse Co-Oximeter. The pulse co-oximeter will non-invasively monitor and record methemoglobin blood levels at 10 second intervals throughout dental treatment. Following a routine oral examination, radiographs, and prophylaxis, subjects assigned to Groups 1 and 2 will be administered local anesthetic for restorative dental treatment. Group 1 subjects will receive 5mg/kg of 4% prilocaine plain and Group 2 subjects will receive 2.5mg/kg of 2% lidocaine with 1:100,000 epinephrine. Group 3 subjects will not receive local anesthetic. The time of local anesthetic administration and baseline methemoglobin blood levels will be recorded. Methemoglobin blood levels will be monitored and recorded throughout the completion of the dental treatment and during recovery from general anesthesia until subject movement precludes any further monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled to undergo comprehensive dental treatment under general anesthesia at the Koppel Special Care Dentistry Center at Loma Linda University School of Dentistry
* ASA I or II health status
* Age greater than 3 years but less than 6 years
* Weigh between 10kg and 25kg

Exclusion Criteria:

* Patient not requiring restorative dental treatment
* Have a BMI less than the 5th percentile or greater than the 95th percentile for their age and gender

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren L Gutenberg, DDS, Study Director — Loma Linda University Department of Pediatric Dentistry; Jung-Wei Chen, DDS, MS, PhD, Principal Investigator — Loma Linda University Department of Pediatric Dentistry
Locations (1):
- Loma Linda University School of Dentistry Koppel Special Care Dentistry Center, Loma Linda, California, United States

REFERENCES:
- [Background] Wright RO, Lewander WJ, Woolf AD. Methemoglobinemia: etiology, pharmacology, and clinical management. Ann Emerg Med. 1999 Nov;34(5):646-56. doi: 10.1016/s0196-0644(99)70167-8. PMID 10533013
- [Background] Ash-Bernal R, Wise R, Wright SM. Acquired methemoglobinemia: a retrospective series of 138 cases at 2 teaching hospitals. Medicine (Baltimore). 2004 Sep;83(5):265-273. doi: 10.1097/01.md.0000141096.00377.3f. PMID 15342970
- [Background] Umbreit J. Methemoglobin--it's not just blue: a concise review. Am J Hematol. 2007 Feb;82(2):134-44. doi: 10.1002/ajh.20738. PMID 16986127
- [Background] Trapp L, Will J. Acquired methemoglobinemia revisited. Dent Clin North Am. 2010 Oct;54(4):665-75. doi: 10.1016/j.cden.2010.06.007. Epub 2010 Aug 7. PMID 20831930
- [Background] Malamed SF. Local anesthetics: dentistry's most important drugs, clinical update 2006. J Calif Dent Assoc. 2006 Dec;34(12):971-6. PMID 17260521
- [Background] Budenz AW. Local anesthetics in dentistry: then and now. J Calif Dent Assoc. 2003 May;31(5):388-96. PMID 12839231
- [Background] Moore PA, Hersh EV. Local anesthetics: pharmacology and toxicity. Dent Clin North Am. 2010 Oct;54(4):587-99. doi: 10.1016/j.cden.2010.06.015. PMID 20831923
- [Background] Bader AM, Concepcion M, Hurley RJ, Arthur GR. Comparison of lidocaine and prilocaine for intravenous regional anesthesia. Anesthesiology. 1988 Sep;69(3):409-12. doi: 10.1097/00000542-198809000-00022. No abstract available. PMID 3415022
- [Background] Vasters FG, Eberhart LH, Koch T, Kranke P, Wulf H, Morin AM. Risk factors for prilocaine-induced methaemoglobinaemia following peripheral regional anaesthesia. Eur J Anaesthesiol. 2006 Sep;23(9):760-5. doi: 10.1017/S0265021506000913. Epub 2006 May 24. PMID 16723054
- [Background] Soeding P, Deppe M, Gehring H. Pulse-oximetric measurement of prilocaine-induced methemoglobinemia in regional anesthesia. Anesth Analg. 2010 Oct;111(4):1065-8. doi: 10.1213/ANE.0b013e3181eb6239. Epub 2010 Aug 12. PMID 20705783
- [Background] Wilburn-Goo D, Lloyd LM. When patients become cyanotic: acquired methemoglobinemia. J Am Dent Assoc. 1999 Jun;130(6):826-31. doi: 10.14219/jada.archive.1999.0306. PMID 10377640
- [Background] Guay J. Methemoglobinemia related to local anesthetics: a summary of 242 episodes. Anesth Analg. 2009 Mar;108(3):837-45. doi: 10.1213/ane.0b013e318187c4b1. PMID 19224791
- [Background] Adams V, Marley J, McCarroll C. Prilocaine induced methaemoglobinaemia in a medically compromised patient. Was this an inevitable consequence of the dose administered? Br Dent J. 2007 Nov 24;203(10):585-7. doi: 10.1038/bdj.2007.1045. PMID 18037845
- [Background] American Academy of Pediatric Dentistry. American Academy of Pediatric Dentistry 2010-2011 Definitions, Oral Health Policies, and Clinical Guidelines: Guidelines on use of local anesthetic for pediatric dental patients. Pediatr Dent 2010;32(6):156-61
- [Background] Yagiela, J. Injectable and topical local anesthetics. In: ADA/PDR guide to dental therapeutics. 5th Edition. Chicago: American Dental Association Publishing Co; 2009 p. 11-2
- [Background] Herdevall BM, Klinge B, Persson L, Huledal G, Abdel-Rehim M. Plasma levels of lidocaine, o-toluidine, and prilocaine after application of 8.5 g Oraqix in patients with generalized periodontitis: effect on blood methemoglobin and tolerability. Acta Odontol Scand. 2003 Aug;61(4):230-4. doi: 10.1080/00016350310004106. PMID 14582591
- [Background] Barker SJ, Curry J, Redford D, Morgan S. Measurement of carboxyhemoglobin and methemoglobin by pulse oximetry: a human volunteer study. Anesthesiology. 2006 Nov;105(5):892-7. doi: 10.1097/00000542-200611000-00008. PMID 17065881
- [Background] Feiner JR, Bickler PE. Improved accuracy of methemoglobin detection by pulse CO-oximetry during hypoxia. Anesth Analg. 2010 Nov;111(5):1160-7. doi: 10.1213/ANE.0b013e3181f46da8. Epub 2010 Sep 14. PMID 20841412
- [Background] Feiner JR, Bickler PE, Mannheimer PD. Accuracy of methemoglobin detection by pulse CO-oximetry during hypoxia. Anesth Analg. 2010 Jul;111(1):143-8. doi: 10.1213/ANE.0b013e3181c91bb6. Epub 2009 Dec 10. PMID 20007731
- [Background] Ash-Bernal R, Brophy GM, Kily D. Acquired methemoglobinemia in the clinical setting: an important health issue revealed. CME Zone Special Report 2006 Nov.
- [Background] Dentsply Pharmaceutical. 4% Citanest Plain Package Insert. York, PA.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients that were greater than 3 years but less than 6 years of age that were scheduled to undergo comprehensive dental rehabilitation under general anesthesia at the Koppel Special Care Dentistry Center at Loma Linda University School of Dentistry were recruited for the study.
Pre-assignment Details: Enrolled participants were excluded prior to group assignment if they had a body mass index (BMI) less than the 5th percentile or greater than the 95th percentile for their age and gender.
Groups:
- Prilocaine: 5mg/kg of 4% prilocaine plain administered via infiltration into multiple sites of the buccal mucosa of the mouth 1 time prior to start of restorative dental treatment
- Lidocaine: 2.5mg/kg of 2% lidocaine with 1:100,000 epinephrine administered via infiltration into multiple sites of the buccal mucosa of the mouth 1 time prior to start of restorative dental treatment
- No Local Anesthetic: No local anesthetic was administered prior to restorative dental treatment-Negative control
Period: Overall Study
Arm/Group | Prilocaine | Lidocaine | No Local Anesthetic
Started | 30 | 30 | 31
Completed | 30 | 30 | 30
Not Completed | 0 | 0 | 1
Not completed — Required Tooth Extraction | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: 1 subject was withdrawn from the no local anesthetic group as the subject required 1 or more dental tooth extractions and required local anesthetic
Groups:
- Total: Total of all reporting groups
Arm/Group | Prilocaine | Lidocaine | No Local Anesthetic | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Continuous [Mean (Standard Deviation); unit: months] | 50.97 (9.84) | 50.77 (10.19) | 50.63 (8.43) | 50.79 (9.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 14 | 45
  Male | 11 | 18 | 16 | 45
Weight Continuous [Mean (Standard Deviation); unit: kilograms] | 17.17 (2.94) | 17.24 (2.78) | 17.19 (2.96) | 17.20 (2.86)
ASA Health Classification [Number; unit: participants]
  I-Healthy patients; no systemic disease | 26 | 25 | 24 | 75
  II-Patients with mild, systemic disease | 4 | 5 | 6 | 15
Body Mass Index Numerical Value [Mean (Standard Deviation); unit: kg/m^2] | 15.62 (1.12) | 15.69 (1.08) | 15.60 (1.03) | 15.64 (1.07)
Body Mass Index Percentile [Number; unit: participants]
  >=5th and <=35th percentiles | 11 | 6 | 6 | 23
  >35th and <=65th percentiles | 6 | 14 | 12 | 32
  >65th and <=95th percentiles | 13 | 10 | 12 | 35
Baseline Methemoglobin Blood Level [Mean (Standard Deviation); unit: percentage] — Methemoglobin blood level recorded non-invasively by the Masimo Radical-7 Pulse Co-Oximeter prior to the administration of local anesthetic or start of restorative dental procedures.
  percentage | 0.82 (0.39) | 0.85 (0.35) | 0.84 (0.43) | 0.83 (0.39)

OUTCOME MEASURES:

1. Primary Outcome: Peak Methemoglobin Blood Levels
Description: The maximum percentage of methemoglobin in blood
Time Frame: Measured at 10 second intervals during dental treatment for an average of 2 hours
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percentage of methemoglobin in blood
Arm/Group | Prilocaine | Lidocaine | No Local Anesthetic
Number analyzed (Participants) | 30 | 30 | 30
percentage of methemoglobin in blood | 3.55 (1.22) | 1.63 (0.52) | 1.60 (0.45)
Statistical Analysis 1: Comparison: Prilocaine vs Lidocaine vs No Local Anesthetic; Null hypothesis: There is no statistically significant difference in peak methemoglobin blood levels following the administration of prilocaine, lidocaine, or no local anesthetic in pre-cooperative children undergoing comprehensive dental rehabilitation under general anesthesia; Test type: Non-Inferiority or Equivalence — Power of 80; p < .001, ANOVA — LSD post hoc test was used for multiple group comparisons. P<.05; LSD post hoc test was used for multiple group comparisons
Statistical Analysis 2: Comparison: Prilocaine vs Lidocaine; LSD post hoc pairwise comparison; Test type: Non-Inferiority or Equivalence — Power of 80; p < .001, Least significant difference post hoc — P<.05
Statistical Analysis 3: Comparison: Prilocaine vs No Local Anesthetic; LSD post hoc pairwise comparison; Test type: Non-Inferiority or Equivalence — Power of 80; p < .001, least significant difference post hoc — P<.05
Statistical Analysis 4: Comparison: Lidocaine vs No Local Anesthetic; LSD post hoc pairwise comparison; Test type: Non-Inferiority or Equivalence — Power of 80; p = .89, Least significant difference post hoc — P<.05

2. Secondary Outcome: Time to Peak Methemoglobin Blood Levels
Description: The length of time between the administration of local anesthetic (Prilocaine and Lidocaine Groups) or start of restorative dental procedures (No local anesthetic Group) and the time at which the maximum methemoglobin blood level is observed.
Time Frame: Measured at 10 second intervals during dental treatment for an average of 2 hours
Population: per protocol
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Prilocaine | Lidocaine | No Local Anesthetic
Number analyzed (Participants) | 30 | 30 | 30
minutes | 62.73 (23.78) | 57.50 (30.67) | 29.50 (20.36)
Statistical Analysis 1: Comparison: Prilocaine vs Lidocaine vs No Local Anesthetic; Null hypothesis: There is no statistically significant difference in the time frame to peak methemoglobin levels following the administration of prilocaine, lidocaine, or no local anesthetic in pre-cooperative children undergoing comprehensive dental rehabilitation under general anesthesia; Test type: Non-Inferiority or Equivalence — Power of 80; p < .001, ANOVA; LSD post hoc test was used for multiple group comparisons
Statistical Analysis 2: Comparison: Prilocaine vs Lidocaine; LSD post hoc pairwise comparison; Test type: Non-Inferiority or Equivalence — Power of 80; p = .43, Least significant difference post hoc — P<.05
Statistical Analysis 3: Comparison: Prilocaine vs No Local Anesthetic; LSD post hoc pairwise comparison; Test type: Non-Inferiority or Equivalence — Power of 80; p < .001, Least significant difference post hoc — P<.05
Statistical Analysis 4: Comparison: Lidocaine vs No Local Anesthetic; LSD post hoc pairwise comparison; Test type: Non-Inferiority or Equivalence — Power of 80; p < .001, Least significant difference post hoc — P<.05

3. Secondary Outcome: Delta Methemoglobin Blood Level
Description: Change in percentage of methemoglobin in blood from baseline level to peak level
Time Frame: From administration of local anesthetic or start of restorative procedures to time at which maximum methemoglobin blood level was documented during dental treatment for an average of 2 hours
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percentage of methemoglobin in blood
Arm/Group | Prilocaine | Lidocaine | No Local Anesthetic
Number analyzed (Participants) | 30 | 30 | 30
percentage of methemoglobin in blood | 2.73 (1.23) | 0.78 (0.44) | 0.76 (0.48)
Statistical Analysis 1: Comparison: Prilocaine vs Lidocaine vs No Local Anesthetic; Null hypothesis: There is no statistically significant difference in delta methemoglobin blood levels following the administration prilocaine, lidocaine, or no local anesthetic in pre-cooperative children undergoing comprehensive dental rehabilitation under general anesthesia; Test type: Non-Inferiority or Equivalence — Power of 80; p < .001, ANOVA — P<.05; LSD post hoc test was used for multiple group comparisons
Statistical Analysis 2: Comparison: Prilocaine vs Lidocaine; LSD post hoc pairwise comparison; Test type: Non-Inferiority or Equivalence — Power of 80; p < .001, Least significant difference post hoc — P<.05
Statistical Analysis 3: Comparison: Prilocaine vs No Local Anesthetic; LSD post hoc pairwise comparison; Test type: Non-Inferiority or Equivalence — Power of 80; p < .001, Least significant difference post hoc — P<.05
Statistical Analysis 4: Comparison: Lidocaine vs No Local Anesthetic; LSD post hoc pairwise comparison; Test type: Non-Inferiority or Equivalence — Power of 80; p = .92, Least significant difference post hoc — P<.05

ADVERSE EVENTS:
Time Frame: Reported adverse events include those that occurred at or after the administration of local anesthetic in the Prilocaine and Lidocaine Groups or the start of restorative dental procedures in the No Local Anesthetic Group.
Arm/Group | Prilocaine | Lidocaine | No Local Anesthetic
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
Did not compare locals anesthetics with equivalent concentrations of epinephrine; unable to control length of time methemoglobin blood levels were monitored as all subjects varied in extent of restorative dental procedures needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes